CLINICAL TRIAL: NCT03696212
Title: Open Label, Single Arm, Phase 1b/2 Study to Evaluate the Safety and Efficacy of Grapiprant (ARY-007) in Combination With Pembrolizumab in Patients With Advanced or Metastatic Post-PD-1/L1 Non-Small Cell Lung Cancer (NSCLC) Adenocarcinoma
Brief Title: Grapiprant (ARY-007) and Pembrolizumab in Patients With Advanced or Metastatic Post-PD-1/L1 NSCLC Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on the totality of the generated combined safety and efficacy data in the interim period, the company decided to terminate the combination study in NSCLC patients. There are no subjects on study drug at this time or in the EOT Follow-up period.
Sponsor: Arrys Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARYS-002; KEYNOTE-888 (Other: MERCK)
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Non-small Cell Lung Cancer Adenocarcinoma
MeSH Terms: interventions — grapiprant; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- grapiprant and pembrolizumab combination (Experimental): Participants will be treated with grapiprant in combination with pembrolizumab.
  Interventions: Drug: grapiprant and pembrolizumab

INTERVENTIONS:
Drug: grapiprant and pembrolizumab — Participants will be administered 21-day cycles of oral grapiprant in combination with IV pembrolizumab
  Other Names: ARYS-007; MK-3475; KEYNOTE-888; IK-007

SUMMARY:
This study will be conducted in adult participants diagnosed with NSCLC who have been previously treated for a minimum of 12 weeks with any PD-1 or PD-L1 checkpoint inhibitor. This is a phase 1b/2, multi-center, open label study designed to assess safety and tolerability of grapiprant in combination with pembrolizumab, to determine the recommended phase 2 dose (RP2D) with pembrolizumab, and to evaluate disease response with grapiprant based on investigator assessments. Pharmacokinetics, pharmacodynamics and response biomarkers will also be assessed.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female adult patients at least 18 years of age on day of signing informed consent
* Histologically confirmed non-small cell lung cancer (NSCLC) adenocarcinoma
* Advanced (stage IIIb) disease that is not amenable to curative intent treatment with concurrent chemoradiation and metastatic (stage IV) patients
* Progressed clinically and/or radiographically per RECIST v1.1 after receiving a PD-1 or PD-L1 antagonist for a minimum of 12 weeks
* Measurable disease per RECIST v1.1
* Disease that can be safely accessed via bronchoscopic, thoracoscopic or percutaneous biopsy for multiple core biopsies and participant is willing to provide tissue from newly obtain biopsies on study in a subgroup of patients
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate organ function
* Highly effective birth control
* Able to swallow and absorb oral tablets

Key Exclusion Criteria:

* Current use of NSAIDs, COX-2 inhibitors
* Known epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), ROS gene alteration
* No history of smoking (≤100 cigarettes lifetime)
* History of severe hypersensitivity reactions to a PD-1/L1 antibody
* Received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment or 5 half-lives, whichever is shorter
* Received prior radiotherapy within 2 weeks of start of study treatment
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Taking strong CYP3A4 or P-glycoprotein inhibitors or inducers
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Known additional malignancy that is progressing or has required active treatment within the past 3 years (with some permitted exceptions)
* Known active CNS metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in past 2 years
* History of pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Recent or current GI ulcer, colitis or non-immune colitis
* Known history of human immunodeficiency virus (HIV) infection, or known active Hepatitis B, or Hepatitis C virus infection
* Has had an allogeneic tissue/solid organ transplant
* Clinically significant (i.e.active) cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of grapiprant in combination with pembrolizumab | Up to 90 days after the end of treatment (average of 7 months)
  Number of incidence, severity, relationship, concomitant medications administered, and duration of treatment emergent adverse events using CTCAE v5.0
Define the recommended phase 2 dose (RP2D) of grapiprant combined with pembrolizumab | Through Cycle 1 (21 days)
  Number, incidence and severity of treatment related adverse events as assessed by CTCAE 5.0
Objective response rate (ORR) | 7 months
  Proportion of participants who achieved PR or better during the study per RECIST 1.1 and iRECIST

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 12 months
  Participants who discontinue treatment without disease progression
Overall survival (OS) | Up to 2 years from start of study drug
  Date of study drug to date of death due to any cause
Duration of treatment (DoT) | 7 months
  Disease response for time of duration on treatment
Disease control rate (DCR) | 7 months
  Percentage of patients who have achieved CR, PR and stable disease
Duration of response (DoR) | Up to 12 months
  Time from documentation of tumor response to disease progression per RECIST and iRECIST 1.1
PK of grapiprant: AUC | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with Cycle 4 (every 42 days) through end of treatment (average of 4 months).
  Area under the plasma concentration-time curve
PK of grapiprant: Cmax | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with Cycle 4 (every 42 days) through end of treatment (average of 4 months).
  Peak serum concentration of grapiprant
Plasma decay half-life (t1/2) | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with Cycle 4 (every 42 days) through end of treatment (average of 4 months).
  Measurement of half-life of grapiprant after dosing
Apparent oral clearance (CL/F) | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with Cycle 4 (every 42 days) through end of treatment (average of 4 months).
  Rate of elimination of the drug from plasma after oral administration
Peak to trough ratio | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with Cycle 4 (every 42 days) through end of treatment (average of 4 months).
  Measure how drug effect is sustained over dose interval
Observed accumulation ratio | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with Cycle 4 (every 42 days) through end of treatment (average of 4 months).
  Relationship between the dosing interval and the rate of elimination for the drug
Pharmacodynamic immune effects in paired tumor biopsies | Predose through cycle 3 (each cycle is 21 days)
  Asses changes in tumor infiltrating helper T cells, cytoxic T cells and regulatory monocyte/macrophages with study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sager, MD, Study Director — Arrys Therapeutics
Locations (6):
- United States (6):
  - Stanford University Medical Center, Stanford, California
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided